CLINICAL TRIAL: NCT01618747
Title: A Single-arm, Open-label, Multicenter, Non-interventional Study to Assess Bevacizumab (Avastin) in Relapsed Glioblastoma
Brief Title: An Observational Study of Avastin (Bevacizumab) in Patients With Glioblastoma Multiforme in First or Second Relapse
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25550
Record Dates: First submitted 2012-06-11; First posted 2012-06-13 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This single-arm, open-label, multicenter, observational study will evaluate the efficacy and safety of Avastin (bevacizumab) in patients with glioblastoma multiforme in first or second relapse. Data will be collected from eligible patients initiated on Avastin treatment according to local label for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients, >/= 18 years of age
* Histologically confirmed glioblastoma multiforme in first or second relapse

Exclusion Criteria:

* Patients not qualifying for Avastin treatment as per local label

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with previously treated glioblastoma multiforme in first or second relapse
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2013-03-15 (Actual); Primary Completion 2015-12-24 (Actual); Study Completion 2015-12-24 (Actual)

PRIMARY OUTCOMES:
Progression-free survival at 6 months | approximately 3 years

SECONDARY OUTCOMES:
Progression-free survival | approximately 3 years
Time to disease progression | approximately 3 years
Duration of objective response | approximately 3 years
Overall survival | approximately 3 years
Safety: Incidence of adverse events | approximately 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- Taiwan (2):
  - Kaohisung
  - Taipei